CLINICAL TRIAL: NCT00548626
Title: EMUNE-07 Evaluation of Multiple Needle Use in EUS-FNA for Pancreatic Cancer
Brief Title: Evaluation of Multiple Needle Use in EUS-FNA for Pancreatic Cancer
Acronym: EMUNE-07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15497A
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Endoscopic Ultrasonography; Fine-Needle Aspiration; Cytopathology
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Needles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients assigned to simple needle group (SN) will be sampled for a total of 6 consecutive FNA passes with a single EUS-FNA needle (only replaced if the needle has a reduced performance). After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.
  Interventions: Procedure: Single needle
- B (Experimental): Patients assigned to multiple needle group (MN) will be sampled for a total of 6 consecutive FNA passes, replacing the needle after every 2 passes. After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.
  Interventions: Procedure: Multiple needle

INTERVENTIONS:
Procedure: Single needle — Patients will be sampled for a total of 6 consecutive FNA passes with a single EUS-FNA needle (only replaced if the needle has a reduced performance). After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.
  Arms: A
Procedure: Multiple needle — Patients will be sampled for a total of 6 consecutive FNA passes, replacing the needle after every 2 passes. After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.
  Arms: B

SUMMARY:
The aim of this study is to evaluate if the early change of needle during EUS-FNA for suspected pancreatic cancer allows an earlier preliminary cytological diagnosis of neoplasia.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial which will recruit patients referred for suspicion of pancreatic mass and indication of EUS-FNA as part of standard of care in the Interventional Endoscopy Unit at the University Of Chicago Medical Center. Basic demographic data will be recorded for each patient. If a pancreatic mass is confirmed in EUS evaluation the patient will be randomized in a 1:1 ratio to either Control group (Single needle) or Investigational group (Multiple Needle). There will be an expert cytopathologist in the exploration room (blinded to the group assignment). Samples obtained through FNA will be prepared onsite either for cytological evaluation by the cytopathologist: each fine needle sample will be expressed by using a 10mL air-filled syringe onto a separate glass slide, and a direct smear will be made by an on-site cytopathologist. Each slide will be air-dried and/or alcohol fixed (95% ethanol), and direct smears will be prepared for immediate interpretation by staining with Diff-quick staining system.

Patients assigned to simple needle group (SN) will be sampled for a total of 6 consecutive FNA passes with a single EUS-FNA needle (only replaced if the needle has a reduced performance). After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.

Patients assigned to multiple needle group (MN) will be sampled for a total of 6 consecutive FNA passes, replacing the needle after every 2 passes. After completing the 6th pass the endoscopist will be informed by the onsite cytopathologist about the preliminary cytological diagnosis.

A cytopathologist (#1) will be present during each EUS-FNA procedure to prepare the slides and determine whether each specimen was adequately cellular. After the procedure, all the cytological samples will be sent to the Pathology department in order to complete the study. A cytopathologist (#2) not present during the procedure will study all the sampling specimens obtained during the EUS-FNA procedure and produce the final and definitive cytopathological diagnosis.

Criteria for pancreatic cancer and benign pancreatic lesions will be defined. Follow-up of all patients to assess early and late complications will be carried out for 30 days after the procedure.

Endpoints:

1. Primary endpoint: Evaluate if the early change of needle during EUS-FNA for suspected pancreatic cancer can reduce the number of passes needed to obtain a preliminary cytological diagnosis of neoplasia. We hypothesized that the number of passes needed using the multiple needles will be significantly less than that using the single needle.
2. Secondary endpoints:

   * Rate of complications related with EUS-FNA
   * Influence of different factors in obtaining a positive cytological result (histological differentiation)

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of pancreatic mass due to previous exam/s (CT, MR, ERCP, US, …) that requires EUS-FNA in order to complete diagnosis
* Age ≥ 18 y/o
* Formal informed consent
* No previous chemotherapy or radiotherapy
* No previous pancreatic surgery

Exclusion Criteria:

* Any patient unable to understand the procedure, nature of the current study, or sign a consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluate if the early change of needle during EUS-FNA for suspected pancreatic cancer can reduce the number of passes needed to obtain a preliminary cytological diagnosis of neoplasia. | October 2007- September 2008

SECONDARY OUTCOMES:
Rate of complications related with EUS-FNA | October 2007- September 2008
Influence of different factors in obtaining a positive cytological result | October 2007- September 2008

CONTACTS AND LOCATIONS:
Overall Officials: Irving Waxman, MD, Principal Investigator — Department of Medicine, University of Chicago Medical Center
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] LeBlanc JK, Ciaccia D, Al-Assi MT, McGrath K, Imperiale T, Tao LC, Vallery S, DeWitt J, Sherman S, Collins E. Optimal number of EUS-guided fine needle passes needed to obtain a correct diagnosis. Gastrointest Endosc. 2004 Apr;59(4):475-81. doi: 10.1016/s0016-5107(03)02863-3. PMID 15044881
- [Background] Wallace MB, Kennedy T, Durkalski V, Eloubeidi MA, Etamad R, Matsuda K, Lewin D, Van Velse A, Hennesey W, Hawes RH, Hoffman BJ. Randomized controlled trial of EUS-guided fine needle aspiration techniques for the detection of malignant lymphadenopathy. Gastrointest Endosc. 2001 Oct;54(4):441-7. doi: 10.1067/mge.2001.117764. PMID 11577304
- [Background] Eloubeidi MA, Tamhane A, Varadarajulu S, Wilcox CM. Frequency of major complications after EUS-guided FNA of solid pancreatic masses: a prospective evaluation. Gastrointest Endosc. 2006 Apr;63(4):622-9. doi: 10.1016/j.gie.2005.05.024. PMID 16564863
- [Background] Eloubeidi MA, Gress FG, Savides TJ, Wiersema MJ, Kochman ML, Ahmad NA, Ginsberg GG, Erickson RA, Dewitt J, Van Dam J, Nickl NJ, Levy MJ, Clain JE, Chak A, Sivak MV Jr, Wong R, Isenberg G, Scheiman JM, Bounds B, Kimmey MB, Saunders MD, Chang KJ, Sharma A, Nguyen P, Lee JG, Edmundowicz SA, Early D, Azar R, Etemad B, Chen YK, Waxman I, Shami V, Catalano MF, Wilcox CM. Acute pancreatitis after EUS-guided FNA of solid pancreatic masses: a pooled analysis from EUS centers in the United States. Gastrointest Endosc. 2004 Sep;60(3):385-9. doi: 10.1016/s0016-5107(04)01714-6. PMID 15332028
- [Background] Harewood GC, Wiersema MJ. Endosonography-guided fine needle aspiration biopsy in the evaluation of pancreatic masses. Am J Gastroenterol. 2002 Jun;97(6):1386-91. doi: 10.1111/j.1572-0241.2002.05777.x. PMID 12094855
- [Background] Eloubeidi MA, Jhala D, Chhieng DC, Chen VK, Eltoum I, Vickers S, Mel Wilcox C, Jhala N. Yield of endoscopic ultrasound-guided fine-needle aspiration biopsy in patients with suspected pancreatic carcinoma. Cancer. 2003 Oct 25;99(5):285-92. doi: 10.1002/cncr.11643. PMID 14579295
- [Background] O'Toole D, Palazzo L, Arotcarena R, Dancour A, Aubert A, Hammel P, Amaris J, Ruszniewski P. Assessment of complications of EUS-guided fine-needle aspiration. Gastrointest Endosc. 2001 Apr;53(4):470-4. doi: 10.1067/mge.2001.112839. PMID 11275888
- [Background] Wiersema MJ, Vilmann P, Giovannini M, Chang KJ, Wiersema LM. Endosonography-guided fine-needle aspiration biopsy: diagnostic accuracy and complication assessment. Gastroenterology. 1997 Apr;112(4):1087-95. doi: 10.1016/s0016-5085(97)70164-1. PMID 9097990
- [Background] Niederhuber JE, Brennan MF, Menck HR. The National Cancer Data Base report on pancreatic cancer. Cancer. 1995 Nov 1;76(9):1671-7. doi: 10.1002/1097-0142(19951101)76:93.0.co;2-r. PMID 8635074
- [Background] Binmoeller KF, Thul R, Rathod V, Henke P, Brand B, Jabusch HC, Soehendra N. Endoscopic ultrasound-guided, 18-gauge, fine needle aspiration biopsy of the pancreas using a 2.8 mm channel convex array echoendoscope. Gastrointest Endosc. 1998 Feb;47(2):121-7. doi: 10.1016/s0016-5107(98)70343-8. PMID 9512275
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Mortensen MB, Pless T, Durup J, Ainsworth AP, Plagborg GJ, Hovendal C. Clinical impact of endoscopic ultrasound-guided fine needle aspiration biopsy in patients with upper gastrointestinal tract malignancies. A prospective study. Endoscopy. 2001 Jun;33(6):478-83. doi: 10.1055/s-2001-14966. PMID 11437039